CLINICAL TRIAL: NCT01388166
Title: ADESPI: Adherence to Spiriva® in Patients With COPD, Measured by Morisky-8 (MMAS-8) Scale, in Routine Medical Practice in Central & Eastern European Region
Brief Title: ADESPI: Adherence to Spiriva® in Patients With COPD (Chronic Obstructive Pulmonary Disease), Measured by Morisky-8 (MMAS-8) Scale, in Routine Medical Practice
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.483
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with COPD
  Interventions: Procedure: Education

INTERVENTIONS:
Procedure: Education — Education

SUMMARY:
The objective of this observational study is to collect and evaluate data on medication adherence of patients on maintenance COPD therapy with long-acting anticholinergic (e.g. Spiriva® delivered by HandiHaler® or Respimat®) using the MMAS-8 questionnaire.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* Male and female ambulatory outpatients being seen in a participating physicians office for routine care,
* Patients with a clinical diagnosis of COPD and already being treated with the maintenance therapy with long-acting anticholinergic (Tiotropium (Spiriva® HandiHaler® or Respimat®) at least 1 month and within product label
* Patient fluent in language of questionnaire and having the cognitive and functional abilities required to fill in the questionnaire alone

Exclusion criteria:

* Uncooperative patients as judged by the physician
* Patients with any conditions excluded as per Country specific package insert
* Patients currently enrolled in any clinical trial which requires a change in medication for their respiratory problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD
Sampling Method: Non-Probability Sample
Enrollment: 1253 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (90):
- Hungary (40):
  - Boehringer Ingelheim Investigational Site 58, Baja
  - Boehringer Ingelheim Investigational Site 85, Békéscsaba
  - Boehringer Ingelheim Investigational Site 61, Budapest
  - Boehringer Ingelheim Investigational Site 62, Budapest
  - Boehringer Ingelheim Investigational Site 63, Budapest
  - Boehringer Ingelheim Investigational Site 66, Budapest
  - Boehringer Ingelheim Investigational Site 67, Budapest
  - Boehringer Ingelheim Investigational Site 68, Budapest
  - Boehringer Ingelheim Investigational Site 89, Budapest
  - Boehringer Ingelheim Investigational Site 90, Budapest
  - Boehringer Ingelheim Investigational Site 55, Cegléd
  - Boehringer Ingelheim Investigational Site 51, Debrecen
  - Boehringer Ingelheim Investigational Site 64, Dunakeszi
  - Boehringer Ingelheim Investigational Site 77, Dunaújváros
  - Boehringer Ingelheim Investigational Site 56, Edelény
  - Boehringer Ingelheim Investigational Site 78, Esztergom
  - Boehringer Ingelheim Investigational Site 86, Érd
  - Boehringer Ingelheim Investigational Site 60, Gyöngyös
  - Boehringer Ingelheim Investigational Site 52, Hajdúnánás
  - Boehringer Ingelheim Investigational Site 81, Kaposvár
  - Boehringer Ingelheim Investigational Site 54, Kecskemét
  - Boehringer Ingelheim Investigational Site 59, Kistokaj
  - Boehringer Ingelheim Investigational Site 71, Komárom
  - Boehringer Ingelheim Investigational Site 74, Komló
  - Boehringer Ingelheim Investigational Site 65, Mátraháza
  - Boehringer Ingelheim Investigational Site 72, Mosonmagyaróvár
  - Boehringer Ingelheim Investigational Site 83, Nyírbátor
  - Boehringer Ingelheim Investigational Site 53, Nyíregyháza
  - Boehringer Ingelheim Investigational Site 88, Nyíregyháza
  - Boehringer Ingelheim Investigational Site 73, Pécs
  - Boehringer Ingelheim Investigational Site 87, Szeged
  - Boehringer Ingelheim Investigational Site 84, Szentes
  - Boehringer Ingelheim Investigational Site 69, Szigetszentmiklós
  - Boehringer Ingelheim Investigational Site 82, Szombathely
  - Boehringer Ingelheim Investigational Site 76, Tapolca
  - Boehringer Ingelheim Investigational Site 79, Tatabánya
  - Boehringer Ingelheim Investigational Site 57, Tiszaújváros
  - Boehringer Ingelheim Investigational Site 70, Törökszentmiklós
  - Boehringer Ingelheim Investigational Site 75, Várpalota
  - Boehringer Ingelheim Investigational Site 80, Zalaegerszeg
- Slovakia (48):
  - Boehringer Ingelheim Investigational Site 29, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 41, Bardejov
  - Boehringer Ingelheim Investigational Site 42, Bardejov
  - Boehringer Ingelheim Investigational Site 32, Bojnice
  - Boehringer Ingelheim Investigational Site 1, Bratislava
  - Boehringer Ingelheim Investigational Site 9, Bratislava
  - Boehringer Ingelheim Investigational Site 45, Čadca
  - Boehringer Ingelheim Investigational Site 28, Galanta
  - Boehringer Ingelheim Investigational Site 17, Gelnica
  - Boehringer Ingelheim Investigational Site 26, Hurbanovo
  - Boehringer Ingelheim Investigational Site 12, Košice
  - Boehringer Ingelheim Investigational Site 13, Košice
  - Boehringer Ingelheim Investigational Site 14, Košice
  - Boehringer Ingelheim Investigational Site 15, Košice
  - Boehringer Ingelheim Investigational Site 16, Košice
  - Boehringer Ingelheim Investigational Site 25, Levice
  - Boehringer Ingelheim Investigational Site 33, Lučenec
  - Boehringer Ingelheim Investigational Site 35, Lučenec
  - Boehringer Ingelheim Investigational Site 36, Lučenec
  - Boehringer Ingelheim Investigational Site 44, Martin
  - Boehringer Ingelheim Investigational Site 38, Michalovce
  - Boehringer Ingelheim Investigational Site 4, Myjava
  - Boehringer Ingelheim Investigational Site 22, Nitra
  - Boehringer Ingelheim Investigational Site 23, Nitra
  - Boehringer Ingelheim Investigational Site 24, Nitra
  - Boehringer Ingelheim Investigational Site 30, Nová Bana
  - Boehringer Ingelheim Investigational Site 48, Nové Mesto N. Váhom
  - Boehringer Ingelheim Investigational Site 19, Nové Zámky
  - Boehringer Ingelheim Investigational Site 20, Nové Zámky
  - Boehringer Ingelheim Investigational Site 21, Nové Zámky
  - Boehringer Ingelheim Investigational Site 5, Piešťany
  - Boehringer Ingelheim Investigational Site 47, Povazská Bystrica
  - Boehringer Ingelheim Investigational Site 39, Prešov
  - Boehringer Ingelheim Investigational Site 40, Prešov
  - Boehringer Ingelheim Investigational Site 31, Prievidza
  - Boehringer Ingelheim Investigational Site 11, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site 34, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site 10, Rožňava
  - Boehringer Ingelheim Investigational Site 2, Senec
  - Boehringer Ingelheim Investigational Site 3, Senica
  - Boehringer Ingelheim Investigational Site 18, Spisská Nová Ves
  - Boehringer Ingelheim Investigational Site 37, Stropkov
  - Boehringer Ingelheim Investigational Site 27, Topoľčany
  - Boehringer Ingelheim Investigational Site 6, Trnava
  - Boehringer Ingelheim Investigational Site 7, Trnava
  - Boehringer Ingelheim Investigational Site 8, Trnava
  - Boehringer Ingelheim Investigational Site 46, Trstená
  - Boehringer Ingelheim Investigational Site 43, Žilina
- Slovenia (2):
  - Boehringer Ingelheim Investigational Site 49, Golnik
  - Boehringer Ingelheim Investigational Site 50, Maribor-Pohorje

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With COPD: Patients with a clinical diagnosis of chronic obstructive pulmonary disease (COPD) being treated with the maintenance therapy with long-acting anticholinergic (Tiotropium) for at least 1 month and within product label.
Period: Overall Study
Arm/Group | Patients With COPD
Started | 1253
Completed | 1194
Not Completed | 59
Not completed — Adverse Event | 16
Not completed — Lost to Follow-up | 30
Not completed — Others than specified above | 13

BASELINE CHARACTERISTICS:
Population: Patients from the Treated Set: This patient set includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment. As it was an inclusion criterion that all patients were treated with Spiriva within the last month, TS consists of all patients involved in the trial.
Arm/Group | Patients With COPD
Number analyzed (Participants) | 1253
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480
  Male | 773

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Morisky Medication Adherence Scale -8 (MMAS-8) Score at the End of the Educational Period After 6 Months From Baseline
Description: The MMAS-8 scale is a recognized indicator of medication adherence, consisting of 8 questions with a sum score ranging between 0 and 8 points. The higher score indicates higher adherence to the prescribed therapy recommendation. It has been agreed that the score of 8 could be categorized as having high adherence, score between 6 and 7 as medium adherence and scores of 5 and less as low adherence. The change is presented as the score on visit 3 minus the score at baseline. Therefore, a positive change score reflects an improvement in the adherence.
Time Frame: Baseline and 6 months
Population: This patient set includes all patients in the TS who have valid MMAS-8 questionnaire results both at baseline and after 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients With COPD
Number analyzed (Participants) | 1168
units on a scale | 0.6 (1.84)
Statistical Analysis 1: Comparison: Patients With COPD; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Mean Change of Morisky Medication Adherence Scale -8 (MMAS-8) Score at the End of the Observational Period After 12 Months From End of Educational Period After 6 Months.
Description: The MMAS-8 scale is a recognized indicator of medication adherence, consisting of 8 questions with a sum score ranging between 0 and 8 points. The higher score indicates higher adherence to the prescribed therapy recommendation. It has been agreed that the score of 8 could be categorized as having high adherence, score between 6 and 7 as medium adherence and scores of 5 and less as low adherence. The change is presented as the score on visit 4 minus the score at visit 3. Therefore, a positive change score reflects an improvement in the adherence.
Time Frame: 6 months and 12 months
Population: This patient set includes all patients in the TS who have valid MMAS-8 questionnaire results after 6 and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients With COPD
Number analyzed (Participants) | 1125
units on a scale | 0.2 (1.46)
Statistical Analysis 1: Comparison: Patients With COPD; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

3. Secondary Outcome: Mean Change of Morisky Medication Adherence Scale -8 (MMAS-8) Score at the End of the Observational Period After 12 Months From Baseline
Description: The MMAS-8 scale is a recognized indicator of medication adherence, consisting of 8 questions with a sum score ranging between 0 and 8 points. The higher score indicates higher adherence to the prescribed therapy recommendation. It has been agreed that the score of 8 could be categorized as having high adherence, score between 6 and 7 as medium adherence and scores of 5 and less as low adherence. The change is presented as the score on visit 4 minus the score at visit 1 (baseline). Therefore, a positive change score reflects an improvement in the adherence.
Time Frame: 12 months and baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients With COPD
Number analyzed (Participants) | 1130
units on a scale | 0.7 (1.82)
Statistical Analysis 1: Comparison: Patients With COPD; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Patients With COPD: Patients with a clinical diagnosis of chronic obstructive pulmonary disease (COPD) being treated with the maintenance therapy with long-acting anticholinergic (Tiotropium) at least 1 months and within product label.
Arm/Group | Patients With COPD
Serious Adverse Events (participants affected / at risk) | 59/1253
Other Adverse Events (participants affected / at risk) | 0/1253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With COPD (N=1253)
Anaemia (Blood and lymphatic system disorders) | 4
Metastases to lymph nodes (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cor pulmonale (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 1
Syncope (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Varices oesophageal (Gastrointestinal disorders) | 1
Death (General disorders) | 4
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Metastases to liver (Hepatobiliary disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 4
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Metastases to bone (Musculoskeletal and connective tissue disorders) | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Vascular encephalopathy (Nervous system disorders) | 1
Amnesia (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Panic disorder (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Ovarian neoplasm (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Lung adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Lung neoplasm (Respiratory, thoracic and mediastinal disorders) | 1
Metastases to lung (Respiratory, thoracic and mediastinal disorders) | 1
Non-small cell lung cancer (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia bacterial (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1
Lung lobectomy (Surgical and medical procedures) | 1
Haemoptysis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.